CLINICAL TRIAL: NCT04739085
Title: Level of Agreement Between Clinical Defocus Curves and the Near and Intermediate Vision Web-based Democritus Digital Acuity Reading Test wDDART: a Comparative Study
Brief Title: Level of Agreement Between Clinical Defocus Curves and the Web-based Democritus Digital Acuity Reading Test wDDART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES1/Th4/21-1-2021
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Presbyopia; Near Vision
Keywords: defocus curves; multifocal IOL implantation; wDDART
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Defocus curve group: The monocular distance visual acuity of each participant' eye is evaluated using trial lenses of -3.00 sph, -2.50 sph, -1.75 sph, and -1.25 sph (added to the best correction for distance), which correspond to the distances of 30 cm, 40 cm, 60 cm, and 80 cm, respectively.
  Interventions: Diagnostic Test: Defocus curves - Monocular distance visual acuity with trial lenses added to the best correction for distance
- wDDART group: The same participants undergo visual acuity test via the web-based digital near vision reading test wDDART at 30 cm, 40 cm, 60 cm and 80 cm, having their best correction for distance.
  Interventions: Diagnostic Test: wDDART - Monocular near visual acuity using the best correction for distance

INTERVENTIONS:
Diagnostic Test: Defocus curves - Monocular distance visual acuity with trial lenses added to the best correction for distance — The monocular distance visual acuity of each participant' eye is evaluated using trial lenses of -3.00 sph, -2.50 sph, -1.75 sph, and -1.25 sph (added to the best correction for distance), which correspond to distances 30 cm, 40 cm, 60 cm and 80 cm, respectively.
  Groups: Defocus curve group
Diagnostic Test: wDDART - Monocular near visual acuity using the best correction for distance — The same participants undergo visual acuity test via the web-based digital near vision reading test wDDART at 30 cm, 40 cm, 60 cm and 80 cm, having their best correction for distance.
  Groups: wDDART group

SUMMARY:
The primary objective of this study is to compare the level of agreement between clinical defocus curves and the web Democritus Digital Acuity Reading Test (wDDART), which is a web-based digital near and intermediate vision reading test.

DETAILED DESCRIPTION:
The 'defocus curve' assessment technique aims to simulate different distances from near to far over which the patient's visual acuity (VA) is evaluated. Defocus curves are created by first measuring best-corrected distance and near VA of the examinee. Then, a series of positive- and negative-powered trial lenses are added to the best-corrected distance visual acuity (BCDVA) of the patient's eye. Viewing through the addition of a minus lens creates divergent light rays with the same refractive effect as bringing the eye chart closer to the viewer. For instance, a -2.50 D lens represents the distance of 40 cm.

The "defocus curve" assessment technique is a method used widely for the assessment of the functional vision range following multifocal intraocular lens (IOL) implantation. Since this method is a simulation of the near vision, it would be ideal if near vision could be evaluated objectively with a near vision chart. However, the conventional printed near vision charts are not available for a variety of reading distances. In addition, the measurement of near VA at different distances with a printed reading chart intended for one predefined distance (e.g. printed chart for 40 cm) and the transformation of the reading score at 40 cm to an equivalent score for the examined distances is impractical in clinical setting.

For this reason, a digital reading test that allows the text calibration for all reading distances could be a practical method for the rapid and ease evaluation of the near VA, especially in patients implanted with multifocal IOLs. The web-based digital near and intermediate vision reading test wDDART offers the ability to estimate VA at different distances with automated measurement of the patient-screen distance.

Therefore, the present study aims to investigate the level of agreement between clinical defocus curves and the web-based digital near and intermediate vision reading test wDDART.

ELIGIBILITY:
Inclusion Criteria:

* Previous cataract lens extraction, age> 40 years, monocular best corrected distance visual acuity > 7/10

Exclusion Criteria:

* Glaucoma, corneal diseases, macular diseases, postoperative opacification of the posterior capsule, former mental diseases

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previous cataract lens extraction will be categorized into the following groups:
  1. Monofocal group
  2. Monovision group (monofocal IOLs bilaterally)
  3. Hybrid monovision group (monofocal IOL in the dominant eye and multifocal IOL in the recessive eye)
  4. Bilateral multifocal group (the same multifocal IOLs bilaterally)
  5. Premium monovision group [bifocal hybrid IOL (Restor +2.50 diopters, Alcon) in the dominant eye and trifocal diffractive IOL (Panoptix, Alcon) in the recessive eye]
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Distance-corrected near visual acuity (DCNVA) at 30 cm via defocus curves | through study completion, 6 months
  The monocular distance visual acuity of each participant's eye is evaluated using a trial lens of -3.00 sph (added to the best correction for distance), which corresponds to the distance of 30 cm
Distance-corrected near visual acuity (DCNVA) at 40 cm via defocus curves | through study completion, 6 months
  The monocular distance visual acuity of each participant's eye is evaluated using a trial lens of -2.50 sph (added to the best correction for distance), which corresponds to the distance of 40 cm
Distance-corrected intermediate visual acuity (DCIVA) at 60 cm via defocus curves | through study completion, 6 months
  The monocular distance visual acuity of each participant's eye is evaluated using a trial lens of -1.75 sph (added to the best correction for distance), which corresponds to the distance of 60 cm
Distance-corrected intermediate visual acuity (DCIVA) at 80 cm via defocus curves | through study completion, 6 months
  The monocular distance visual acuity of each participant's eye is evaluated using a trial lens of -1.25 sph (added to the best correction for distance), which corresponds to the distance of 80 cm
Distance-corrected near visual acuity (DCNVA) at 30 cm via wDDART | through study completion, 6 months
  The monocular near (30 cm) visual acuity of each participant's eye is evaluated using the best correction for distance
Distance-corrected near visual acuity (DCNVA) at 40 cm via wDDART | through study completion, 6 months
  The monocular near (40 cm) visual acuity of each participant's eye is evaluated using the best correction for distance
Distance-corrected intermediate visual acuity (DCIVA) at 60 cm via wDDART | through study completion, 6 months
  The monocular intermediate (60 cm) visual acuity of each participant's eye is evaluated using the best correction for distance
Distance-corrected intermediate visual acuity (DCIVA) at 80 cm via wDDART | through study completion, 6 months
  The monocular intermediate (80 cm) visual acuity of each participant's eye is evaluated using the best correction for distance

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Background] Labiris G, Panagiotopoulou EK, Chatzimichael E, Tzinava M, Mataftsi A, Delibasis K. Introduction of a digital near-vision reading test for normal and low vision adults: development and validation. Eye Vis (Lond). 2020 Oct 22;7:51. doi: 10.1186/s40662-020-00216-0. eCollection 2020. PMID 33102611